CLINICAL TRIAL: NCT01331707
Title: DUrable Polymer-based STent CHallenge of Promus Element Versus ReSolute Integrity (DUTCH PEERS): Randomized Multicenter Trial in All Comers Population Treated Within Eastern NeThErlands-2 (TWENTE-2)
Brief Title: DUrable Polymer-based STent CHallenge of Promus Element Versus ReSolute Integrity in an All Comers Population
Acronym: DUTCH PEERS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation of Cardiovascular Research and Education Enschede (Other)
Responsible Party: Principal Investigator, prof. C. von Birgelen, Professor C. von Birgelen, Thorax Centrum Twente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUTCH PEERS; NTR2413 (Registry Identifier: Dutch trial register entry)
Record Dates: First submitted 2011-03-30; First posted 2011-04-08 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Acute Coronary Syndrome; Angina Pectoris; Angina, Unstable; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis
Keywords: drug-eluting stent; Zotarolimus; Everolimus; all comers population; target vessel failure; coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris; Angina, Unstable; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Promus Element (Active Comparator)
  Interventions: Device: Promus Element (Everolimus-eluting stent)
- Resolute Integrity (Active Comparator)
  Interventions: Device: Resolute Integrity (Zotarolimus-eluting stent)

INTERVENTIONS:
Device: Resolute Integrity (Zotarolimus-eluting stent) — Third generation drug-eluting stent
  Arms: Resolute Integrity
Device: Promus Element (Everolimus-eluting stent) — Third generation drug-eluting stent
  Arms: Promus Element

SUMMARY:
The introduction of drug-eluting stents (DES) in the treatment of coronary artery disease has led to a significant reduction in morbidity but there are further demands on DES performance. Such demands are an optimized performance in very challenging coronary lesions; third generation DES were developed in an effort to further improve DES performance in such challenging lesions. Two CE-certified third generation DES (Resolute Integrity and Promus Element stents) are currently available; there are no data that indicate an advantage of one of these DES over the other.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years;
* Coronary artery disease and lesion(s) eligible for treatment with drug eluting stents according to clinical guidelines and/or the operators' judgement;
* Patient is willing and able to cooperate with study procedures and required follow-up visits; and patient has been informed and agrees on the participation by signing an EC approved written informed consent.

Exclusion Criteria:

* Participation in another randomized drug or device study before reaching primary endpoint;
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period;
* Intolerance to a P2Y12 receptor antagonist that results in the patient's inability to adhere to dual-antiplatelet therapy, or intolerance to aspirin, heparin, or components of the two DES examined;
* Known pregnancy;
* Life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1811 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF): a composite of Cardiac death, Target vessel related Myocardial Infarction and Clinically driven repeated target vessel revascularization | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Medisch Centrum Alkmaar, Alkmaar
  - Hospital Rijnstate, Arnhem
  - Scheper Hospital, Emmen
  - Thoraxcentrum Twente, Enschede

REFERENCES:
- [Derived] Pinxterhuis TH, Ploumen EH, Doggen CJM, van Vliet D, Kok MM, Zocca P, Hartmann M, van Houwelingen KG, Stoel MG, de Man FHAF, Linssen GCM, von Birgelen C. Sex and age-specific 10-year mortality after coronary stenting: an analysis of two randomized trials. Eur Heart J Open. 2025 Jan 29;5(1):oeaf006. doi: 10.1093/ehjopen/oeaf006. eCollection 2025 Jan. PMID 39959922
- [Derived] Pinxterhuis TH, Ploumen EH, van Vliet D, Gert van Houwelingen K, Stoel MG, de Man FH, Hartmann M, Zocca P, Linssen GC, Geelkerken RH, Doggen CJ, von Birgelen C. Ten-year mortality after treating obstructive coronary atherosclerosis with contemporary stents in patients with or without concomitant peripheral arterial disease. Atherosclerosis. 2024 May;392:117488. doi: 10.1016/j.atherosclerosis.2024.117488. Epub 2024 Mar 26. PMID 38598970
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Hartmann M, Linssen GCM, von Birgelen C. Impact of premature coronary artery disease on adverse event risk following first percutaneous coronary intervention. Front Cardiovasc Med. 2023 Sep 7;10:1160201. doi: 10.3389/fcvm.2023.1160201. eCollection 2023. PMID 37745109
- [Derived] Pinxterhuis TH, Ploumen EH, Doggen CJM, Hartmann M, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Linssen GCM, von Birgelen C. First myocardial infarction in patients with premature coronary artery disease: insights into patient characteristics and outcome after treatment with contemporary stents. Eur Heart J Acute Cardiovasc Care. 2023 Nov 16;12(11):774-781. doi: 10.1093/ehjacc/zuad098. PMID 37619976
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Stoel MG, Linssen GCM, Geelkerken RH, von Birgelen C. Outcome after percutaneous coronary intervention with contemporary stents in patients with concomitant peripheral arterial disease: A patient-level pooled analysis of four randomized trials. Atherosclerosis. 2022 Aug;355:52-59. doi: 10.1016/j.atherosclerosis.2022.05.002. Epub 2022 May 20. PMID 35641327
- [Derived] Zocca P, Kok MM, Tandjung K, Danse PW, Jessurun GAJ, Hautvast RWM, van Houwelingen KG, Stoel MG, Schramm AR, Tjon Joe Gin RM, de Man FHAF, Hartmann M, Louwerenburg JHW, Linssen GCM, Lowik MM, Doggen CJM, von Birgelen C. 5-Year Outcome Following Randomized Treatment of All-Comers With Zotarolimus-Eluting Resolute Integrity and Everolimus-Eluting PROMUS Element Coronary Stents: Final Report of the DUTCH PEERS (TWENTE II) Trial. JACC Cardiovasc Interv. 2018 Mar 12;11(5):462-469. doi: 10.1016/j.jcin.2017.11.031. PMID 29519378
- [Derived] van der Heijden LC, Kok MM, Lowik MM, Danse PW, Jessurun GAJ, Hartmann M, Stoel MG, van Houwelingen KG, Hautvast RWM, Linssen GC, Doggen CJM, von Birgelen C. Three-Year Clinical Outcome of Patients with Coronary Disease and Increased Event Risk Treated with Newer-Generation Drug-Eluting Stents: From the Randomized DUTCH PEERS Trial. Cardiology. 2017;137(4):207-217. doi: 10.1159/000464320. Epub 2017 Apr 27. PMID 28445871
- [Derived] van der Heijden LC, Kok MM, Danse PW, Schramm AR, Hartmann M, Lowik MM, Linssen GC, Stoel MG, Doggen CJ, von Birgelen C. Small-vessel treatment with contemporary newer-generation drug-eluting coronary stents in all-comers: Insights from 2-year DUTCH PEERS (TWENTE II) randomized trial. Am Heart J. 2016 Jun;176:28-35. doi: 10.1016/j.ahj.2016.02.020. Epub 2016 Mar 17. PMID 27264217
- [Derived] von Birgelen C, Sen H, Lam MK, Danse PW, Jessurun GA, Hautvast RW, van Houwelingen GK, Schramm AR, Gin RM, Louwerenburg JW, de Man FH, Stoel MG, Lowik MM, Linssen GC, Said SA, Nienhuis MB, Verhorst PM, Basalus MW, Doggen CJ, Tandjung K. Third-generation zotarolimus-eluting and everolimus-eluting stents in all-comer patients requiring a percutaneous coronary intervention (DUTCH PEERS): a randomised, single-blind, multicentre, non-inferiority trial. Lancet. 2014 Feb 1;383(9915):413-23. doi: 10.1016/S0140-6736(13)62037-1. Epub 2013 Oct 31. PMID 24183564
- [Derived] Tandjung K, Basalus MW, Sen H, Jessurun GA, Danse PW, Stoel M, Linssen GC, Derks A, van Loenhout TT, Nienhuis MB, Hautvast RW, von Birgelen C. DUrable polymer-based sTent CHallenge of Promus ElemEnt versus ReSolute integrity (DUTCH PEERS): rationale and study design of a randomized multicenter trial in a Dutch all-comers population. Am Heart J. 2012 Apr;163(4):557-62. doi: 10.1016/j.ahj.2012.02.001. PMID 22520520